CLINICAL TRIAL: NCT01939197
Title: A Multipart, Open-label Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/Ritonavir With and Without Dasabuvir Coadministered With and Without Ribavirin in Adults With Genotype 1 or 4 Chronic Hepatitis C Virus Infection and Human Immunodeficiency Virus, Type 1 Coinfection (TURQUOISE-I)
Brief Title: A Multipart, Open-label Study to Evaluate the Safety and Efficacy of ABT-450/r/ABT-267 With and Without ABT-333 Coadministered With and Without Ribavirin in Adult With Genotype 1 or 4 Hepatitis C Virus (HCV) Infection and Human Immunodeficiency Virus, Type 1 Coinfection
Acronym: TURQUOISE-I
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-004; 2012-005143-24 (EudraCT Number)
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C Virus Infection; Human Immunodeficiency Virus Infection; Chronic Hepatitis C; Compensated Cirrhosis and Non-cirrhotics
Keywords: HCV Genotype 4; Interferon-Free; Hepatitis C Genotype 1; Compensated Cirrhosis; Hepatitis C Genotype 4; HCV / HIV coinfection; Cirrhotic; Hepatitis C; HIV-1; HCV Genotype 1
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome; Hepatitis C, Chronic; HIV Infections | interventions — ombitasvir; paritaprevir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- ARM A (Experimental): ABT-450/r/ABT-267 and ABT-333 coadministered with ribavirin (RBV) for 12 weeks for participants receiving atazanavir once-daily or raltegravir twice-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: ribavirin
- ARM B (Experimental): ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 24 weeks for participants receiving atazanavir once-daily or raltegravir twice-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: ribavirin
- ARM C (Experimental): ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving darunavir once-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: ribavirin
- ARM D (Experimental): ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving darunavir twice-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: ribavirin
- ARM E (Experimental): ABT-450/r/ABT-267 and ABT-333 for 12 weeks for noncirrhotic (at screening) GT1b-infected participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333
- ARM F (Experimental): ABT-450/r/ABT-267 and ABT-333 for 12 weeks for cirrhotic (at screening) GT1b-infected sofosbuvir-naive participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333
- ARM G (Experimental): ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for cirrhotic (at screening) GT1b-infected sofosbuvir-naive participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: ribavirin
- ARM H (Experimental): ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for cirrhotic (at screening) GT1b-infected sofosbuvir-experienced participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: ribavirin
- ARM I (Experimental): ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for noncirrhotic (at screening) GT1a-infected participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: ribavirin
- ARM J (Experimental): ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 24 weeks for cirrhotic (at screening) GT1a-infected participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: ribavirin
- ARM K (Experimental): ABT-450/r/ABT-267 coadministered with RBV for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily, dolutegravir once-daily or twice-daily, darunavir once-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ribavirin
- ARM L (Experimental): ABT-450/r/ABT-267 coadministered with RBV for 24 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily, dolutegravir once-daily or twice-daily, darunavir once-daily
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ribavirin

INTERVENTIONS:
Drug: ABT-450/r/ABT-267 — tablet
  Other Names: ombitasvir/paritaprevir/ritonavir; ombitasvir also known as ABT-267; paritaprevir also known as ABT-450
Drug: ABT-333 — tablet
  Other Names: Dasabuvir
  Arms: ARM A; ARM B; ARM C; ARM D; ARM E; ARM F; ARM G; ARM H; ARM I; ARM J
Drug: ribavirin — tablet
  Arms: ARM A; ARM B; ARM C; ARM D; ARM G; ARM H; ARM I; ARM J; ARM K; ARM L

SUMMARY:
The primary objectives of this study are to assess the safety of ABT-450/r/ABT-267 with and without ABT-333 coadministered with and without ribavirin (RBV) for 12 and 24 weeks in HCV GT1- or 4-infected participants with HIV-1 coinfection and to evaluate the percentage of subjects achieving HCV ribonucleic acid (RNA) < lower limit of quantification (LLOQ) 12 weeks following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection at screening defined as: positive anti-HCV antibodies (Ab) at screening and HCV RNA > 1,000 IU/mL at screening.
* Plasma HIV-1 RNA < 40 copies/mL during screening using Abbott RealTime HIV-1 assay.
* On a stable qualifying HIV-1 antiretroviral therapy regimen.

Exclusion Criteria:

* Positive test result at screening for hepatitis B surface antigen.
* Evidence of HCV genotype other than genotype 1 or genotype 4 during screening.
* Receipt of any other investigational or commercially available anti-HCV agents (for example, telaprevir, boceprevir, simeprevir, daclatasvir and ledipasvir) with the exception of interferon (including pegylated-interferon alfa-2a or alfa-2b), sofosbuvir and ribavirin.
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive ABT-450, ABT-267, ABT-333, ritonavir or ribavirin.
* Chronic human immunodeficiency virus, type 2 (HIV-2) infection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2013-08-30; Primary Completion 2016-07-21 (Actual); Study Completion 2016-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolando Viani, MD, Study Director — AbbVie

REFERENCES:
- [Background] Sulkowski MS, Eron JJ, Wyles D, Trinh R, Lalezari J, Wang C, Slim J, Bhatti L, Gathe J, Ruane PJ, Elion R, Bredeek F, Brennan R, Blick G, Khatri A, Gibbons K, Hu YB, Fredrick L, Schnell G, Pilot-Matias T, Tripathi R, Da Silva-Tillmann B, McGovern B, Campbell AL, Podsadecki T. Ombitasvir, paritaprevir co-dosed with ritonavir, dasabuvir, and ribavirin for hepatitis C in patients co-infected with HIV-1: a randomized trial. JAMA. 2015 Mar 24-31;313(12):1223-31. doi: 10.1001/jama.2015.1328. PMID 25706092
- [Derived] Kwo PY, Poordad F, Asatryan A, Wang S, Wyles DL, Hassanein T, Felizarta F, Sulkowski MS, Gane E, Maliakkal B, Overcash JS, Gordon SC, Muir AJ, Aguilar H, Agarwal K, Dore GJ, Lin CW, Liu R, Lovell SS, Ng TI, Kort J, Mensa FJ. Glecaprevir and pibrentasvir yield high response rates in patients with HCV genotype 1-6 without cirrhosis. J Hepatol. 2017 Aug;67(2):263-271. doi: 10.1016/j.jhep.2017.03.039. Epub 2017 Apr 13. PMID 28412293
- [Derived] King JR, Khatri A, Trinh R, Viani RM, Ding B, Zha J, Menon R. Pharmacokinetic Evaluation of Darunavir Administered Once or Twice Daily in Combination with Ritonavir or the Three-Direct-Acting Antiviral Regimen of Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir in Adults Coinfected with Hepatitis C and Human Immunodeficiency Viruses. Antimicrob Agents Chemother. 2017 Jan 24;61(2):e02135-16. doi: 10.1128/AAC.02135-16. Print 2017 Feb. PMID 27919899
- [Derived] Saeed S, Strumpf EC, Walmsley SL, Rollet-Kurhajec K, Pick N, Martel-Laferriere V, Hull M, Gill MJ, Cox J, Cooper C, Klein MB; Canadian Co-Infection Cohort Study; Cohen J, Conway B, Cooper C, Cote P, Cox J, Gill J, Haider S, Harris M, Haase D, Hull M, Montaner J, Moodie E, Pick N, Rachlis A, Rouleau D, Sandre R, Tyndall JM, Vachon ML, Walmsley S, Wong D. How Generalizable Are the Results From Trials of Direct Antiviral Agents to People Coinfected With HIV/HCV in the Real World? Clin Infect Dis. 2016 Apr 1;62(7):919-926. doi: 10.1093/cid/civ1222. Epub 2016 Jan 6. PMID 26743093
- See also: This clinical study may be evaluating a usage that is not currently FDA-approved. Please see US Prescribing Information for approved uses. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 2 was not designed to test different treatments on the same subject population. Rather, the arms in Part 2 represent subpopulations with different baseline characteristics (hepatitis C virus [HCV] genotype [GT], cirrhotic status, prior HCV therapy experience). Arms F and G were randomized to regimens without and with ribavirin, respectively.
Pre-assignment Details: In Part 2, participants in Arms E, F, H, I, J all had GT1 infection and received 1 consistent treatment regimen based on label recommendations; they were therefore combined and named the "GT1 Analysis Group."
Groups:
- Part 1a: Arm A: ABT-450/r/ABT-267 and ABT-333 coadministered with ribavirin (RBV) for 12 weeks for participants receiving atazanavir once-daily or raltegravir twice-daily
- Part 1a: Arm B: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 24 weeks for participants receiving atazanavir once-daily or raltegravir twice-daily
- Part 1b: Arm C: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving darunavir once-daily
- Part 1b: Arm D: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving darunavir twice-daily
- Part 2: GT1 Analysis Group: Participants with HCV genotype (GT)1a or GT1b at screening in Arms E, F, H, I, J (no participants enrolled in Arm H) Arm E: ABT-450/r/ABT-267 and ABT-333 for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily Arm F: ABT-450/r/ABT-267 and ABT-333 for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily Arm I: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily Arm J: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 24 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
- Part 2: Arm G: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
- GT4 Analysis Group: Participants with HCV GT4 at screening in Arms K and L (no participants enrolled in Arm L).
  Arm K: ABT-450/r/ABT-267 coadministered with RBV for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily, dolutegravir once-daily or twice-daily, darunavir once-daily
Period: Overall Study
Arm/Group | Part 1a: Arm A | Part 1a: Arm B | Part 1b: Arm C | Part 1b: Arm D | Part 2: GT1 Analysis Group | Part 2: Arm G | GT4 Analysis Group
Started | 31 | 32 | 10 | 12 | 200 | 5 | 28
Completed | 30 | 31 | 10 | 11 | 196 | 4 | 26
Not Completed | 1 | 1 | 0 | 1 | 4 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Part 1a: Arm A: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving atazanavir once-daily or raltegravir twice-daily
- Part 2: GT1 Analysis Group: Participants with HCV GT1a or GT1b at screening in Arms E, F, H, I, J (no participants enrolled in Arm H) Arm E: ABT-450/r/ABT-267 and ABT-333 for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily Arm F: ABT-450/r/ABT-267 and ABT-333 for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily Arm I: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily Arm J: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 24 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
- Part 2: GT4 Analysis Group: Arm K: ABT-450/r/ABT-267 coadministered with RBV for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily, dolutegravir once-daily or twice-daily, darunavir once-daily Arm L: no participants enrolled
- Total: Total of all reporting groups
Arm/Group | Part 1a: Arm A | Part 1a: Arm B | Part 1b: Arm C | Part 1b: Arm D | Part 2: GT1 Analysis Group | Part 2: Arm G | Part 2: GT4 Analysis Group | Total
Number analyzed (Participants) | 31 | 32 | 10 | 12 | 200 | 5 | 28 | 318
Age, Customized [Count of Participants; unit: Participants]
  Age Group: < 55 years | 23 | 20 | 5 | 8 | 145 | 2 | 24 | 227
  Age Group: ≥ 55 years | 8 | 12 | 5 | 4 | 55 | 3 | 4 | 91
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 3 | 44 | 1 | 2 | 57
  Male | 29 | 29 | 8 | 9 | 156 | 4 | 26 | 261

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in GT1 Analysis Group 1 in Part 2 Achieving Sustained Virologic Response 12 Weeks Post-Treatment (SVR12)
Description: SVR12 is defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (< LLOQ) 12 weeks after the last dose of study drug without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window. The 95% confidence interval (CI) is calculated using the Wilson score method for binomial distribution.
  The primary efficacy endpoint was the non-inferiority of the percentage of participants in the GT1 Analysis Group in Part 2 achieving SVR12 compared to the historical SVR12 rate for sofosbuvir plus ribavirin (a non-inferiority threshold of the lower bound of the 95% CI of 74%).
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat population: Part 2 randomized or enrolled participants who received at least 1 dose of study drug. Imputation applied; participants with missing HCV RNA data after imputation were counted as failures. The primary efficacy endpoint analysis was based on subjects in the GT 1 Analysis Group in Part 2 containing Arms E, F, H, I, and J.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: GT1 Analysis Group
Number analyzed (Participants) | 200
percentage of participants | 97.0 [93.6 to 98.6]
Statistical Analysis 1: Comparison: Part 2: GT1 Analysis Group; Test type: Non-Inferiority — The primary efficacy endpoint was the non-inferiority of the percentage of participants in the GT1 Analysis Group in Part 2 achieving SVR12 compared to the historical SVR12 rate for sofosbuvir plus ribavirin (a non-inferiority threshold of the lower bound of the 95% CI of 74%); The historical SVR rate, as reported in the PHOTON-1 study, for sofosbuvir and RBV in HCV/HIV-1 coinfected adults is 76% (87/114) with a 95% confidence interval of (67%, 84%). Reference: Sulkowski MS, Naggie S, Lalezari J, et al. Sofosbuvir and ribavirin for hepatitis C in patients with HIV coinfection. JAMA. 2014;312(4):353-61

2. Secondary Outcome: Percentage of Participants in Part 1a Achieving SVR12
Description: SVR12 is defined as plasma HCV RNA < LLOQ 12 weeks after the last dose of study drug without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window. The 95% CI is calculated using the Wilson score method for binomial distribution.
Time Frame: 12 weeks after last dose of study drug
Population: Intent-to-treat population: Part 1a randomized participants who received at least 1 dose of study drug. Imputation applied; participants with missing HCV RNA data after imputation were counted as failures.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1a: Arm A | Part 1a: Arm B
Number analyzed (Participants) | 31 | 32
percentage of participants | 93.5 [79.3 to 98.2] | 90.6 [75.8 to 96.8]
Statistical Analysis 1: Comparison: Part 1a: Arm A vs Part 1a: Arm B; Test type: Other; p = 1.000, Fisher Exact

3. Secondary Outcome: Percentage of Participants in Part 1b Achieving SVR12
Description: as for outcome 2
Time Frame: 12 weeks after last dose of study drug
Population: Intent-to-treat population: Part 1b randomized participants who received at least 1 dose of study drug. Imputation applied; participants with missing HCV RNA data after imputation were counted as failures.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1b: Total: Arm C: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving darunavir once-daily
  Arm D: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving darunavir twice-daily
Arm/Group | Part 1b: Arm C | Part 1b: Arm D | Part 1b: Total
Number analyzed (Participants) | 10 | 12 | 22
percentage of participants | 100 [72.2 to 100.0] | 100 [75.8 to 100.0] | 100 [85.1 to 100.0]
Statistical Analysis 1: Comparison: Part 1b: Arm C vs Part 1b: Arm D; Test type: Other; The Fisher exact test was performed as prespecified on the SAP but the p-value couldn't be calculated because SVR12 rates in both arms were 100%, hence p-value appeared as "not available."

4. Secondary Outcome: Percentage of Participants in Arm F and Arm G of Part 2 Achieving SVR12
Description: as for outcome 2
Time Frame: 12 weeks after last dose of study drug
Population: Intent-to-treat population: Part 2 randomized or enrolled participants who received at least 1 dose of study drug. Imputation applied; participants with missing HCV RNA data after imputation were counted as failures.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2: Arm F: ABT-450/r/ABT-267 and ABT-333 for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
Arm/Group | Part 2: Arm F | Part 2: Arm G
Number analyzed (Participants) | 4 | 5
percentage of participants | 75.0 [30.1 to 95.4] | 80.0 [37.6 to 96.4]

5. Secondary Outcome: Percentage of Participants With GT4 HCV in Part 2 Achieving SVR12, by Arm and Overall
Description: as for outcome 2
Time Frame: 12 weeks after last dose of study drug
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2: Arm K: ABT-450/r/ABT-267 coadministered with RBV for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily, dolutegravir once-daily or twice-daily, darunavir once-daily
Arm/Group | Part 2: GT4 Analysis Group | Part 2: Arm K
Number analyzed (Participants) | 28 | 28
percentage of participants | 96.4 [82.3 to 99.4] | 96.4 [82.3 to 99.4]

6. Secondary Outcome: Percentage of Participants in Part 1a With On-Treatment HCV Virologic Failure During the Treatment Period
Description: Percentage of participants with on-treatment HCV virologic failure during the treatment period for each arm in Part 1a. Virologic failure is defined as confirmed quantifiable HCV RNA among participants with previously unquantifiable HCV RNA during treatment.
Time Frame: up to 12 or 24 weeks, based on treatment duration
Population: Intent-to-treat population: Part 1a randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1a: Arm A | Part 1a: Arm B
Number analyzed (Participants) | 31 | 32
percentage of participants | 0 [0.0 to 11.0] | 3.1 [0.6 to 15.7]

7. Secondary Outcome: Percentage of Participants in Part 1b With On-Treatment HCV Virologic Failure During the Treatment Period
Description: Percentage of participants with on-treatment HCV virologic failure during the treatment period for each arm and overall in Part 1b. Virologic failure is defined as confirmed quantifiable HCV RNA among participants with previously unquantifiable HCV RNA during treatment.
Time Frame: up to 12 weeks
Population: Intent-to-treat population: Part 1b randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1b: Arm C | Part 1b: Arm D | Part 1b: Total
Number analyzed (Participants) | 10 | 12 | 22
percentage of participants | 0 [0.0 to 27.8] | 0 [0.0 to 24.2] | 0 [0.0 to 14.9]

8. Secondary Outcome: Percentage of Participants in Part 2 With On-Treatment HCV Virologic Failure During the Treatment Period
Description: Percentage of participants with on-treatment HCV virologic failure during the treatment period for arms in Part 2. Virologic failure is defined as confirmed quantifiable HCV RNA among participants with previously unquantifiable HCV RNA during treatment.
Time Frame: up to 12 or 24 weeks, based on treatment duration
Population: Intent-to-treat population: Part 2 randomized or enrolled participants in the GT1 analysis group (and its composing arms) and GT4 analysis group who received at least 1 dose of study drug. Due to a label change after study start that no longer recommended the Arm G treatment regimen to GT1b cirrhotic subjects, Arm G data was not analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2: Arm E; Part 2: Arm F: ABT-450/r/ABT-267 and ABT-333 for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
- Part 2: Arm I: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
- Part 2: Arm J: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 24 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily
- Part 2: GT4 Analysis Group: ABT-450/r/ABT-267 coadministered with RBV for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily, dolutegravir once-daily or twice-daily, darunavir once-daily Arm L: no participants enrolled
- Group 2: Arm K: ABT-450/r/ABT-267 coadministered with RBV for 12 weeks for participants receiving any of the following: atazanavir once-daily, raltegravir twice-daily, dolutegravir once-daily or twice-daily, darunavir once-daily
Arm/Group | Part 2: GT1 Analysis Group | Part 2: Arm E | Part 2: Arm F | Part 2: Arm I | Part 2: Arm J | Part 2: GT4 Analysis Group | Group 2: Arm K
Number analyzed (Participants) | 200 | 42 | 4 | 135 | 19 | 28 | 28
percentage of participants | 0.5 [0.1 to 2.8] | 0 [0.0 to 8.4] | 25.0 [4.6 to 69.9] | 0 [0.0 to 2.8] | 0 [0.0 to 16.8] | 0 [0.0 to 12.1] | 0 [0.0 to 12.1]

9. Secondary Outcome: Percentage of Participants in Part 1a With Relapse12
Description: Percentage of participants who experienced Relapse12 among participants who completed treatment with HCV RNA < LLOQ at final treatment visit and had at least one post-treatment HCV RNA value. Relapse12 is defined as confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after last actual dose of study drug (up to and including the SVR12 assessment time point) for a participant with HCV RNA < LLOQ at final treatment visit who completed treatment and had post-treatment data. Completion of treatment is defined as study drug duration ≥ 77 days for Arm A and ≥ 154 days for Arm B. The 95% CI is calculated using Wilson score method for the binomial distribution.
Time Frame: up to 12 or 24 weeks, based on treatment duration, after the last actual dose of study drug
Population: Intent-to-treat population: Part 1a randomized participants who received at least 1 dose of study drug and who completed treatment with HCV RNA < LLOQ at final treatment visit and had at least one post-treatment HCV RNA value.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1a: Arm A | Part 1a: Arm B
Number analyzed (Participants) | 30 | 31
percentage of participants | 3.3 [0.6 to 16.7] | 0 [0.0 to 11.0]

10. Secondary Outcome: Percentage of Participants in Part 1b With Relapse12 for Each Arm and Overall
Description: Percentage of participants who experienced Relapse12 among participants who completed treatment with HCV RNA < LLOQ at final treatment visit and had at least one post-treatment HCV RNA value. Relapse12 is defined as confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after last actual dose of study drug (up to and including the SVR12 assessment time point) for a participant with HCV RNA < LLOQ at final treatment visit who completed treatment and had post-treatment data. Completion of treatment is defined as study drug duration ≥ 77 days for Arm C and Arm D. The 95% CI is calculated using Wilson score method for the binomial distribution.
Time Frame: up to 12 weeks after the last actual dose of study drug
Population: Intent-to-treat population: all Part 1b randomized participants who received at least 1 dose of study drug and who completed treatment with HCV RNA < LLOQ at final treatment visit and had at least one post-treatment HCV RNA value.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1b: Arm C | Part 1b: Arm D | Part 1b: Total
Number analyzed (Participants) | 10 | 12 | 22
percentage of participants | 0 [0.0 to 27.8] | 0 [0.0 to 24.2] | 0 [0.0 to 14.9]

11. Secondary Outcome: Percentage of Participants in Part 2 With Relapse12
Description: Percentage of participants who experienced Relapse12 among those who completed treatment with HCV RNA < LLOQ at final treatment visit and had ≥1 post-treatment HCV RNA value. Relapse12=confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after last actual dose of study drug (up to and including the SVR12 window) for a participant with HCV RNA < LLOQ at final treatment visit who completed treatment and had post-treatment data, excluding reinfection. Completion of treatment=study drug duration ≥ 77 days for participants who received 12 weeks of treatment and ≥154 days for participants who received 24 weeks of treatment. HCV reinfection=confirmed HCV RNA ≥ LLOQ after the end of treatment in a subject who had HCV RNA < LLOQ at final treatment visit, along with the post-treatment detection of a different HCV genotype, subtype, or clade compared with baseline, as determined by phylogenetic analysis. The 95% CI is calculated using Wilson score method for the binomial distribution.
Time Frame: up to 12 or 24 weeks, based on treatment duration, after the last actual dose of study drug
Population: Intent-to-treat population: Part 2 randomized or enrolled participants in the GT1 analysis group (and its composing arms) and GT4 analysis group who received ≥1 dose of study drug, who completed treatment with HCV RNA < LLOQ at final treatment visit, and had ≥1 post-treatment HCV RNA value. Arm G data was not analyzed (see Outcome Measure 8).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: GT1 Analysis Group | Part 2: Arm E | Part 2: Arm F | Part 2: Arm I | Part 2: Arm J | Part 2: GT4 Analysis Group | Group 2: Arm K
Number analyzed (Participants) | 192 | 42 | 3 | 131 | 16 | 27 | 27
percentage of participants | 0.5 [0.1 to 2.9] | 0 [0.0 to 8.4] | 0 [0.0 to 56.1] | 0.8 [0.1 to 4.2] | 0 [0.0 to 19.4] | 0 [0.0 to 12.5] | 0 [0.0 to 12.5]

12. Secondary Outcome: Percentage of Participants in Part 1a With Plasma HIV-1 RNA Suppression at End of Treatment and 12 Weeks Post-Treatment
Description: HIV virologic success was defined as HIV-1 RNA suppression (HIV-1 RNA value < 40 copies/mL).
Time Frame: End of treatment: HIV Week 12 window for 12-weeks of treatment (Treatment Day 71 - 98) or HIV Week 24 window (Treatment Day 155 - 182) for 24-weeks of treatment. Post-Treatment Week 12 (PTW12): HIV PTW12 window (Post-Treatment Day 57 - 126)
Population: Intent-to-treat population: Part 1a randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1a: Arm A | Part 1a: Arm B
Number analyzed (Participants) | 31 | 32
percentage of participants
  End of Treatment | 93.5 [79.3 to 98.2] | 90.6 [75.8 to 96.8]
  Post-Treatment Week 12 | 96.8 [83.8 to 99.4] | 93.8 [79.9 to 98.3]

13. Secondary Outcome: Percentage of Participants in Part 1b With Plasma HIV-1 RNA Suppression at End of Treatment and 12 Weeks Post-Treatment
Description: HIV virologic success was defined as HIV-1 RNA suppression (HIV-1 RNA value < 40 copies/mL).
Time Frame: End of treatment: HIV Week 12 window (Treatment Day 78 - 98). PTW12: HIV PTW12 window (Post-Treatment Day 57 - 126)
Population: Intent-to-treat population: Part 1b randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1b Total: Arm C: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving darunavir once-daily
  Arm D: ABT-450/r/ABT-267 and ABT-333 coadministered with RBV for 12 weeks for participants receiving darunavir twice-daily
Arm/Group | Part 1b: Arm C | Part 1b: Arm D | Part 1b Total
Number analyzed (Participants) | 10 | 12 | 22
percentage of participants
  End of Treatment | 100 [72.2 to 100.0] | 83.3 [55.2 to 95.3] | 90.9 [72.2 to 97.5]
  Post-Treatment Week 12 | 100 [72.2 to 100.0] | 75.0 [46.8 to 91.1] | 86.4 [66.7 to 95.3]

14. Secondary Outcome: Percentage of Participants in Part 2 With Plasma HIV-1 RNA Suppression at End of Treatment and 12 Weeks Post-Treatment
Description: HIV virologic success was defined as HIV-1 RNA suppression (HIV-1 RNA value < 40 copies/mL).
Time Frame: End of treatment: HIV Week 12 window for 12-weeks of treatment (Treatment Day 71 - 98) or HIV Week 24 window (Treatment Day 155 - 182) for 24-weeks of treatment. PTW12: HIV PTW12 window (Post-Treatment Day 57 - 126)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: GT1 Analysis Group | Part 2: Arm E | Part 2: Arm F | Part 2: Arm I | Part 2: Arm J | Part 2: GT4 Analysis Group | Group 2: Arm K
Number analyzed (Participants) | 200 | 42 | 4 | 135 | 19 | 28 | 28
percentage of participants
  End of Treatment | 89 [83.9 to 92.6] | 90.5 [77.9 to 96.2] | 100 [51.0 to 100.0] | 89.6 [83.3 to 93.7] | 78.9 [56.7 to 91.5] | 85.7 [68.5 to 94.3] | 85.7 [68.5 to 94.3]
  Post-Treatment Week 12 | 93 [88.6 to 95.8] | 97.6 [87.7 to 99.6] | 100 [51.0 to 100.0] | 91.9 [86.0 to 95.4] | 89.5 [68.6 to 97.1] | 92.9 [77.4 to 98.0] | 92.9 [77.4 to 98.0]

ADVERSE EVENTS:
Time Frame: Protocol-related treatment-emergent adverse events were collected from the first dose of study drug through end of treatment Week 12 and Week 24; treatment-emergent serious adverse events were collected from the first dose of study drug until post treatment Day 30.
Description: A protocol-related event is defined as any event with onset or worsening reported by a participant from the first dose of study drug until 30 days have elapsed following discontinuation of study drug administration. Events were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Part 1a: Arm A | Part 1a: Arm B | Part 1b: Arm C | Part 1b: Arm D | Part 2: Arm E | Part 2: Arm F | Part 2: Arm G | Part 2: Arm I | Part 2: Arm J | Part 2: Arm K
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32 | 0/10 | 1/12 | 1/42 | 0/4 | 0/5 | 6/135 | 2/19 | 1/28
Other Adverse Events (participants affected / at risk) | 28/31 | 27/32 | 10/10 | 10/12 | 23/42 | 3/4 | 4/5 | 109/135 | 18/19 | 23/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1a: Arm A (N=31) | Part 1a: Arm B (N=32) | Part 1b: Arm C (N=10) | Part 1b: Arm D (N=12) | Part 2: Arm E (N=42) | Part 2: Arm F (N=4) | Part 2: Arm G (N=5) | Part 2: Arm I (N=135) | Part 2: Arm J (N=19) | Part 2: Arm K (N=28)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PERICARDITIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
RECTAL PERFORATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DRUG DEPENDENCE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
URETEROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1a: Arm A (N=31) | Part 1a: Arm B (N=32) | Part 1b: Arm C (N=10) | Part 1b: Arm D (N=12) | Part 2: Arm E (N=42) | Part 2: Arm F (N=4) | Part 2: Arm G (N=5) | Part 2: Arm I (N=135) | Part 2: Arm J (N=19) | Part 2: Arm K (N=28)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 3 | 1 | 2 | 0 | 0 | 1 | 6 | 1 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BLEPHAROSPASM (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DRY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
EYE DISCHARGE (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EYE PRURITUS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
EYELID HAEMATOMA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
EYELID PTOSIS (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OCULAR DISCOMFORT (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OCULAR HYPERAEMIA (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
OCULAR ICTERUS (Eye disorders) | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 5 | 0 | 3
APHTHOUS ULCER (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 7 | 2 | 2
DIARRHOEA (Gastrointestinal disorders) | 1 | 4 | 1 | 2 | 4 | 1 | 0 | 26 | 1 | 1
DIVERTICULUM (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
DYSPEPSIA (Gastrointestinal disorders) | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 10 | 0 | 3
FAECES SOFT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 5 | 6 | 2 | 2 | 3 | 1 | 0 | 34 | 4 | 5
ORAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 11 | 1 | 3
ASTHENIA (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 13 | 2 | 3
CHEST PAIN (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
EARLY SATIETY (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 18 | 12 | 5 | 4 | 2 | 0 | 0 | 40 | 6 | 5
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
PAIN (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 0 | 0
PERIPHERAL SWELLING (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2
TEMPERATURE INTOLERANCE (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
TENDERNESS (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VESSEL PUNCTURE SITE BRUISE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 4 | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0 | 1
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
ACUTE SINUSITIS (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 6 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
HERPES ZOSTER OTICUS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 12 | 4 | 4
ORAL HERPES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
PYURIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RHINITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2
SECONDARY SYPHILIS (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 5 | 1 | 0 | 3 | 0 | 0 | 12 | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 6 | 2 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 3 | 0 | 1 | 4 | 0 | 0 | 0 | 13 | 6 | 4
WEIGHT DECREASED (Investigations) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 3 | 0 | 1 | 3 | 1 | 1
GOUT (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 3 | 1 | 0 | 5 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1 | 2 | 0 | 0 | 6 | 3 | 1
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 10 | 2 | 1
HEADACHE (Nervous system disorders) | 6 | 4 | 2 | 1 | 2 | 0 | 1 | 22 | 4 | 5
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
NEURALGIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
SINUS HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
AFFECT LABILITY (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0
AGITATION (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 11 | 1 | 2
DEPRESSED MOOD (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 1
INSOMNIA (Psychiatric disorders) | 5 | 7 | 1 | 0 | 3 | 0 | 1 | 25 | 2 | 2
IRRITABILITY (Psychiatric disorders) | 3 | 3 | 3 | 2 | 0 | 1 | 0 | 7 | 2 | 1
LIBIDO INCREASED (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
STRESS (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2 | 0 | 1 | 0 | 0 | 7 | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 8 | 2 | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 1 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 6 | 2 | 0 | 1 | 1 | 1 | 0 | 18 | 2 | 1
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 6 | 2 | 1
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 4 | 0 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.